CLINICAL TRIAL: NCT03500549
Title: A Phase III, Randomized, Multi-Center, Open-Label, Active-Comparator Controlled Study to Evaluate the Efficacy and Safety of APL-2 in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Study to Evaluate the Efficacy and Safety of APL-2 in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APL2-302
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — pegcetacoplan; eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegcetacoplan (Experimental): 1080 mg pegcetacoplan administered subcutaneously twice-weekly or every three days.
  Interventions: Drug: Pegcetacoplan; Drug: Soliris
- Eculizumab (Active Comparator): Complement (C5) Inhibitor.
  Interventions: Drug: Pegcetacoplan; Drug: Soliris

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) Inhibitor
  Other Names: APL-2
Drug: Soliris — Complement (C5) Inhibitor

SUMMARY:
Evaluation of the Efficacy and Safety of APL-2 in Patients with Paroxysmal Nocturnal Hemoglobinuria

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Primary diagnosis of PNH confirmed by high-sensitivity flow cytometry
* On treatment with eculizumab. Dose of eculizumab must have been stable for at least 3 months prior to the Screening Visit
* Hb <10.5 g/dL at the Screening Visit
* Absolute reticulocyte count > 1.0x ULN at the Screening Visit
* Platelet count of >50,000/mm3 at the Screening Visit
* Absolute neutrophil count >500/mm3 at the Screening Visit
* Vaccination against Neisseria meningitides types A, C, W, Y and B, Streptococcus pneumoniae and Haemophilus influenzae Type B (Hib) either within 2 years prior to Day 1 dosing, or within 14 days after starting treatment with APL-2. Unless documented evidence exists that subjects are non-responders to vaccination as evidenced by titers or display titer levels within acceptable local limits
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test at the Screening and Day -28 Visit (Run-in Period) and must agree to use protocol defined methods of contraception for the duration of the study and 90 days after their last dose of study drug
* Males must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study and 90 days after their last dose of study drug
* Willing and able to give informed consent
* Willing and able to self-administer APL-2 (administration by caregiver will be allowed)
* Have a body mass index (BMI) ≤35.0 kg/m2

Exclusion Criteria:

* Active bacterial infection that has not resolved within 14 week of Day -28 (first dose of APL-2)
* Receiving iron, folic acid, vitamin B12 and EPO, unless the dose is stable, in the 4 weeks prior to Screening
* Hereditary complement deficiency
* History of bone marrow transplantation
* History or presence of hypersensitivity or idiosyncratic reaction to compounds related to the investigational product or SC administration
* Participation in any other investigational drug trial or exposure to other investigational agent within 30 days or 5 half-lives (whichever is longer)
* Currently breast-feeding women
* Inability to cooperate or any condition that, in the opinion of the investigator, could increase the subject's risk of participating in the study or confound the outcome of the study

This study includes cardiac safety evaluations. The following cardiac eligibility criteria are necessary to avoid confounding the cardiac safety outcomes:

* History or family history of Long QT Syndrome or torsade de pointes, unexplained syncope, syncope from an uncorrected cardiac etiology, or family history of sudden death
* Myocardial infarction, CABG, coronary or cerebral artery stenting and /or angioplasty, stroke, cardiac surgery, or hospitalization for congestive heart failure within 3 months or greater than Class 2 Angina Pectoris or NYHA Heart Failure Class >2
* QTcF > 470 ms, PR > 280 ms
* Mobitz II 2nd degree AV Block, 2:1 AV Block, High Grade AV Block, or Complete Heart Block unless the patient has an implanted pacemaker or implantable cardiac defibrillator (ICD) with backup pacing capabilities
* Receiving Class 1 or Class 3 antiarrhythmic agents, or arsenic, methadone, ondansetron or pentamidine at screening
* Receiving any other QTc-prolonging drugs (see Appendix 4 in Section 19.4), at a stable dose for less than 3 weeks prior to dosing
* Receiving prophylactic ciprofloxacin, erythromycin or azithromycin for less than one week prior to the first dose of study medication (must have a repeat screening ECG after one week of prophylactic antibiotics with QTcF < 470 ms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (19):
  - University of Southern California, Los Angeles, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Denver Health, Denver, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Lakes Research, Miami Lakes, Florida
  - Mid Florida Hematology and Oncology, Orange City, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Cancer & Blood Specialists, East Setauket, New York
  - New York Cancer & Blood Specialists, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Good Samaritan Hospital, Corvallis, Oregon
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - HOPE Cancer Center of East Texas, Tyler, Texas
- Royal Melbourne Hospital, Melbourne, Victoria, Australia
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Vlaams-Brabant
  - AZ Delta Campus Wilgenstraat, Roeselare, West-Vlaanderen
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Toronto General Hospital, Toronto, Ontario
- France (8):
  - Centre Hospitalier Annecy Genevois, Annecy
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre Hospitalier Universitaire de Lille, Lille
  - Institut Paoli-Calmettes Marseille, Marseille
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
- Germany (4):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- Japan (8):
  - Japanese Red Cross Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - Japanese Red Cross Nagoya Daini Hospital, Showa-ku, Aichi-ken
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Shinshu University Hospital, Matsumoto, Nagano
  - Okayama University Hospital, Okayama, Okayama-ken
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Kinan Hospital, Tanabe, Wakayama
- Russia (3):
  - Pavlov First Saint Petersburg State Medical University of Russian Ministry of Health, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Institution of Health Care of Tyumen Region, Tyumen
- South Korea (3):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Chungnam National University Hospital, Daejeon
  - Samsung Medical Center, Seoul
- Spain (2):
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario Politécnico La Fe, Valencia
- St. James' Institute of Oncology, Leeds Teaching Hospitals, Leeds, United Kingdom

REFERENCES:
- [Derived] de Castro C, Kelly RJ, Griffin M, Patriquin CJ, Mulherin B, Hochsmann B, Selvaratnam V, Wong RSM, Hillmen P, Horneff R, Uchendu UO, Zhang Y, Surova E, Szamosi J, de Latour RP. Efficacy and Safety Maintained up to 3 Years in Adults with Paroxysmal Nocturnal Hemoglobinuria Receiving Pegcetacoplan. Adv Ther. 2025 Sep;42(9):4641-4658. doi: 10.1007/s12325-025-03310-8. Epub 2025 Jul 28. PMID 40720060
- [Derived] de Latour RP, Kulasekararaj A, Dingli D, Wilson K, Wojciechowski P, Hakimi Z, Nazir J, Czech B, Hillmen P, Szer J. Anchored Indirect Treatment Comparison Finds Comparable Effects of Pegcetacoplan and Iptacopan in Paroxysmal Nocturnal Haemoglobinuria. Eur J Haematol. 2025 Aug;115(2):125-133. doi: 10.1111/ejh.14422. Epub 2025 Apr 25. PMID 40285403
- [Derived] Panse J, Daguindau N, Okuyama S, Peffault de Latour R, Schafhausen P, Straetmans N, Al-Adhami M, Persson E, Wong RSM. Improvements in hematologic markers and decreases in fatigue with pegcetacoplan for patients with paroxysmal nocturnal hemoglobinuria and mild or moderate anemia (hemoglobin >/=10 g/dL) who had received eculizumab or were naive to complement inhibitors. PLoS One. 2024 Jul 29;19(7):e0306407. doi: 10.1371/journal.pone.0306407. eCollection 2024. PMID 39079163
- [Derived] Mulherin BP, Yeh M, Al-Adhami M, Dingli D. Normalization of Hemoglobin, Lactate Dehydrogenase, and Fatigue in Patients with Paroxysmal Nocturnal Hemoglobinuria Treated with Pegcetacoplan. Drugs R D. 2024 Jun;24(2):169-177. doi: 10.1007/s40268-024-00463-9. Epub 2024 May 10. PMID 38727860
- [Derived] Peffault de Latour R, Griffin M, Kelly RJ, Szer J, de Castro C, Horneff R, Tan L, Yeh M, Panse J. Hemolysis events in the phase 3 PEGASUS study of pegcetacoplan in patients with paroxysmal nocturnal hemoglobinuria. Blood Adv. 2024 Jun 11;8(11):2718-2725. doi: 10.1182/bloodadvances.2024012672. PMID 38593241
- [Derived] Sharma V, Koprivnikar J, Drago K, Savage J, Bachelor A. Injection Site Reactions with Long-Term Pegcetacoplan Use in Patients with Paroxysmal Nocturnal Hemoglobinuria: A Brief Report. Adv Ther. 2023 Nov;40(11):5115-5129. doi: 10.1007/s12325-023-02653-4. Epub 2023 Sep 14. PMID 37707673
- [Derived] de Latour RP, Szer J, Weitz IC, Roth A, Hochsmann B, Panse J, Usuki K, Griffin M, Kiladjian JJ, de Castro CM, Nishimori H, Ajayi T, Al-Adhami M, Deschatelets P, Francois C, Grossi F, Risitano AM, Hillmen P. Pegcetacoplan versus eculizumab in patients with paroxysmal nocturnal haemoglobinuria (PEGASUS): 48-week follow-up of a randomised, open-label, phase 3, active-comparator, controlled trial. Lancet Haematol. 2022 Sep;9(9):e648-e659. doi: 10.1016/S2352-3026(22)00210-1. PMID 36055332
- [Derived] Cella D, Sarda SP, Hsieh R, Fishman J, Hakimi Z, Hoffman K, Al-Adhami M, Nazir J, Cutts K, Lenderking WR. Changes in hemoglobin and clinical outcomes drive improvements in fatigue, quality of life, and physical function in patients with paroxysmal nocturnal hemoglobinuria: post hoc analyses from the phase III PEGASUS study. Ann Hematol. 2022 Sep;101(9):1905-1914. doi: 10.1007/s00277-022-04887-8. Epub 2022 Jul 23. PMID 35869984
- [Derived] Hakimi Z, Wilson K, McAughey E, Pochopien M, Wojciechowski P, Toumi M, Knight C, Sarda SP, Patel N, Wiseman C, de Castro NP, Nazir J, Kelly RJ. The cost-effectiveness, of pegcetacoplan compared with ravulizumab for the treatment of paroxysmal nocturnal hemoglobinuria, in a UK setting. J Comp Eff Res. 2022 Sep;11(13):969-985. doi: 10.2217/cer-2022-0076. Epub 2022 Jul 7. PMID 35796199
- [Derived] Bhak RH, Mody-Patel N, Baver SB, Kunzweiler C, Yee CW, Sundaresan S, Swartz N, Duh MS, Krishnan S, Sarda SP. Comparative effectiveness of pegcetacoplan versus ravulizumab in patients with paroxysmal nocturnal hemoglobinuria previously treated with eculizumab: a matching-adjusted indirect comparison. Curr Med Res Opin. 2021 Nov;37(11):1913-1923. doi: 10.1080/03007995.2021.1971182. Epub 2021 Sep 3. PMID 34445916
- [Derived] Hillmen P, Szer J, Weitz I, Roth A, Hochsmann B, Panse J, Usuki K, Griffin M, Kiladjian JJ, de Castro C, Nishimori H, Tan L, Hamdani M, Deschatelets P, Francois C, Grossi F, Ajayi T, Risitano A, Peffault de Latour R. Pegcetacoplan versus Eculizumab in Paroxysmal Nocturnal Hemoglobinuria. N Engl J Med. 2021 Mar 18;384(11):1028-1037. doi: 10.1056/NEJMoa2029073. PMID 33730455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, randomized, multicenter, open-label, active-comparator controlled study evaluated the efficacy and safety of pegcetacoplan (APL-2) in subjects with paroxysmal nocturnal hemoglobinuria who had received treatment with eculizumab (Soliris®) in the past.
Pre-assignment Details: The treatment period of the study consisted of 3 parts: a 4-week run-in period, a 16-week randomized controlled period (RCP), and a 32-week open-label period. Of the 102 subjects screened, 80 subjects met all the inclusion criteria and none of the exclusion criteria and entered the run-in period. Randomization was stratified by the number of packed red blood cell (PRBC) transfusions within the 12 months prior to Day -28 and platelet count at screening.
Groups:
- Pegcetacoplan to Pegcetacoplan: During the 4-week run-in period (Day -28 to ≤Day 1) all subjects received twice-weekly subcutaneous (SC) doses of pegcetacoplan 1080 milligrams (mg) in addition to their current dosage of eculizumab treatment. On Day 1, the subjects were randomized to receive monotherapy with SC infusions of pegcetacoplan 1080 mg twice-weekly or every 3 days up to the end of the open-label period (Week 48).
- Eculizumab to Pegcetacoplan: During the 4-week run-in period (Day -28 to ≤Day 1) all subjects received twice-weekly SC doses of pegcetacoplan 1080 mg in addition to their current dosage of eculizumab treatment. On Day 1, the subjects were randomized to receive monotherapy with their pre-screening stable dose of eculizumab via intravenous infusion every 2 weeks up to the end of the RCP (Week 16). Subjects then entered the open-label run-in period where they received pegcetacoplan 1080 mg twice-weekly in addition to eculizumab for 4 weeks (Week 17 to Week 20) before crossing over to monotherapy with SC infusions of pegcetacoplan 1080 mg twice-weekly or every 3 days up to the end of the open-label period (Week 48).
Period: Run-in Period (Day -28 to ≤Day 1)
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Started | 41 | 39
Completed | 41 | 39
Not Completed | 0 | 0
Period: RCP (Day 1 - Week 16)
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Started | 41 | 39
Completed (Completed treatment at Week 16 analysis.) | 38 | 39
Not Completed | 3 | 0
Not completed — Adverse Event | 3 | 0
Period: Open-label Period (Week 17 to Week 48)
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Started | 38 | 39
Completed (Completed treatment at Week 48 analysis.) | 35 | 32
Not Completed | 3 | 7
Not completed — Adverse Event | 3 | 7

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) set included all randomized subjects.
Groups:
- Pegcetacoplan to Pegcetacoplan: During the 4-week run-in period (Day -28 to ≤Day 1) all subjects received twice-weekly SC doses of pegcetacoplan 1080 mg in addition to their current dosage of eculizumab treatment. On Day 1, the subjects were randomized to receive monotherapy with SC infusions of pegcetacoplan 1080 mg twice-weekly or every 3 days up to the end of the open-label period (Week 48).
- Total: Total of all reporting groups
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 63
  >=65 years | 10 | 7 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 14 | 17 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 29 | 32 | 61
  Unknown or Not Reported | 10 | 6 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 7 | 12
  Black or African American | 2 | 0 | 2
  White | 24 | 25 | 49
  Other | 0 | 1 | 1
  Not Reported | 10 | 6 | 16
Number of transfusions in the last 12 months prior to Day -28 [Count of Participants; unit: Participants]
  < 4 | 20 | 16 | 36
  ≥ 4 | 21 | 23 | 44
Platelet count at screening [Count of Participants; unit: Participants]
  <100,000 (count/mm^3) | 12 | 9 | 21
  ≥100,000 (count/mm^3) | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Least Squares (LS) Mean Change From Baseline to Week 16 in Hemoglobin (Hb) Level During the RCP
Description: Baseline was the average of measurements recorded before taking the first dose of pegcetacoplan, which included local and central laboratory values during the screening period. Analysis excluded data before the RCP and was censored for transfusions.
Time Frame: Baseline and Week 16
Population: The ITT set included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter (g/dL)
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
Grams per deciliter (g/dL) | 2.37 (0.363) | -1.47 (0.666)
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Superiority — The primary endpoint analysis was a between-treatment-group comparison using a mixed effect model for repeated measures (MMRM). The difference between pegcetacoplan and eculizumab LS mean Hb changes from Baseline at Week 16 was calculated along with its 2-sided 95% confidence interval (CI) and associated P-value from the MMRM model for the ITT set, censored for transfusions; p < 0.0001, MMRM — Superiority was tested at the 5% level. MMRM includes treatment + baseline value + analysis visit + strata + analysis visit × treatment, where strata is the combination of randomization stratification factors; LS mean difference = 3.84, 95% CI 2-sided [2.33 to 5.34]

2. Secondary Outcome: Percentage of Subjects Who Did Not Require a Transfusion (Transfusion Avoidance) During the RCP
Description: Subjects who experienced more than 1 transfusion during the RCP are only counted once. Subjects who did not have a transfusion but withdrew before Week 16 were considered as having a transfusion in the analysis of transfusion avoidance.
Time Frame: Day 1 to Week 16
Population: The ITT set included all randomized subjects.
Measure: Number; unit: Percentage of subjects
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
Percentage of subjects | 85.4 | 15.4
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Non-Inferiority — Analysis was based on prespecified non-inferiority margins (NIM) and non-inferiority was achieved if the lower confidence limit or upper confidence limit of the 95% CI of the treatment difference met the prespecified NIM of -20%. Stratified Cochran-Mantel Haenszel (CMH) chi-square test was used for treatment comparison and the 95% CI for difference in percentage between treatments is constructed using the stratified (Miettinen-Nurminen) method; p < 0.0001, Miettinen-Nurminen — Non-inferiority was tested at the 2.5% level; Risk Difference (RD) = 0.6253, 95% CI 2-sided [0.4830 to 0.7677]

3. Secondary Outcome: LS Mean Change From Baseline to Week 16 in Absolute Reticulocyte Count (ARC) During the RCP
Description: Baseline was the average of available measurements recorded from central laboratory before taking the first dose of pegcetacoplan. Analysis excluded data before the RCP and was censored for transfusions.
Time Frame: Baseline and Week 16
Population: The ITT set included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: 10^9 cells/ liter (L)
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
10^9 cells/ liter (L) | -135.82 (6.543) | 27.79 (11.859)
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Non-Inferiority — Analysis was based on prespecified NIM and non-inferiority was achieved if the lower confidence limit or upper confidence limit of the 95% CI of the treatment difference met the prespecified NIM of 10; p < 0.0001, MMRM — Non-inferiority was tested at the 2.5% level. MMRM includes treatment + baseline value + analysis visit + strata + analysis visit × treatment, where strata is the combination of randomization stratification factors; LS mean difference = -163.61, 95% CI 2-sided [-189.91 to -137.30]

4. Secondary Outcome: LS Mean Change From Baseline to Week 16 in Lactate Dehydrogenase (LDH) Level During the RCP
Description: as for outcome 3
Time Frame: Baseline and Week 16
Population: The ITT set included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Units (U)/L
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
Units (U)/L | -14.76 (42.708) | -10.12 (71.025)
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Non-Inferiority — Analysis was based on prespecified NIM and non-inferiority was achieved if the lower confidence limit or upper confidence limit of the 95% CI of the treatment difference met the prespecified NIM of 20; p = 0.9557, MMRM — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -4.63, 95% CI 2-sided [-181.30 to 172.04]

5. Secondary Outcome: LS Mean Change From Baseline to Week 16 in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Scale Score During the RCP
Description: The FACIT-fatigue scale version 4 is a 13-item Likert scaled instrument where the subject was presented with 13 statements and asked to indicate their response as it applied to the past 7 days. The 5 possible responses were 'Not at all' (0), 'A little bit (1), 'Somewhat' (2), 'Quite a bit' (3) and 'Very much' (4). With 13 statements the total score had a range of 0 to 52. A higher score corresponds to a higher quality of life (QoL). Baseline was the last available, nonmissing observation before taking the first dose of pegcetacoplan. Data collected after transfusion is excluded from analysis.
Time Frame: Baseline and Week 16
Population: The ITT set included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
Score on a scale | 9.22 (1.607) | -2.65 (2.821)
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Other — Non-inferiority was not assessed because of the prespecified hierarchical testing. Analysis was a between-treatment-group comparison using an MMRM. The difference between pegcetacoplan and eculizumab LS mean changes from Baseline at Week 16 was calculated along with its 2-sided 95% CI and associated P-value from the MMRM model for the ITT set, censored for transfusions; p = 0.0005, MMRM — MRMM includes treatment + baseline value + analysis visit + strata + analysis visit × treatment, where strata is the combination of randomization stratification factors; LS mean difference = 11.87, 95% CI 2-sided [5.49 to 18.25]

6. Secondary Outcome: Percentage of Subjects Who Achieved a Hb Response in the Absence of Transfusions at Week 16
Description: Hb response was defined as an increase of at least 1 g/dL in Hb from Baseline at Week 16. Baseline was the average of measurements recorded before taking the first dose of pegcetacoplan, which included local and central laboratory values during the screening period. Analysis excluded data before the RCP and was censored for transfusions.
Time Frame: Baseline and Week 16
Population: The ITT set included all randomized subjects.
Measure: Number; unit: Percentage of subjects
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
Percentage of subjects | 75.6 | 0.0
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Other — Stratified CMH chi-square test was used for treatment comparison and the 95% CI for difference in percentage between treatments is constructed using the stratified Miettinen-Nurminen method; Difference in percentage = 0.6745, 95% CI 2-sided [0.5452 to 0.8039] — The difference in percentage and 95% CI is calculated based on stratified Miettinen-Nurminen method stratified by randomization factor so it it is not a direct difference of two reporting groups

7. Secondary Outcome: Percentage of Subjects Who Achieved Reticulocyte Normalization in the Absence of Transfusions at Week 16
Description: Reticulocyte normalization was defined as the ARC being below the upper limit of the gender-specific normal range at Week 16, censored for transfusions. Subjects who received a transfusion between Day 1 and Week 16 or withdrew without providing efficacy data at Week 16 were classified as nonresponders.
Time Frame: Week 16
Population: The ITT set includes all randomized subjects.
Measure: Number; unit: Percentage of subjects
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
Percentage of subjects | 78.0 | 2.6
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Other — [test comment as in outcome 6, analysis 1]; Difference in percentage = 0.6639, 95% CI 2-sided [0.5309 to 0.7968] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Percentage of Subjects Who Achieved Hb Normalization in the Absence of Transfusions at Week 16
Description: Hb normalization was defined as the Hb level being above the lower limit of the normal range at Week 16, censored for transfusions. Subjects who received a transfusion between Day 1 and Week 16 or withdrew without providing efficacy data at Week 16 are classified as nonnormalization.
Time Frame: Week 16
Population: The ITT set included all randomized subjects.
Measure: Number; unit: Percentage of subjects
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
Percentage of subjects | 34.1 | 0.0
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Other — [test comment as in outcome 6, analysis 1]; Difference in percentage = 0.3043, 95% CI 2-sided [0.1493 to 0.4593] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: LS Mean Change From Baseline to Week 16 in Indirect Bilirubin Level During the RCP
Description: as for outcome 3
Time Frame: Baseline and Week 16
Population: The ITT set included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Micromole (μmol)/L
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
Micromole (μmol)/L | -17.78 (2.727) | 4.15 (4.477)
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Other — Analysis was a between-treatment-group comparison using an MMRM. The difference between pegcetacoplan and eculizumab LS mean changes from Baseline at Week 16 was calculated along with its 2-sided 95% CI and associated P-value from the MMRM model for the ITT set, censored for transfusions; p = 0.0002, MMRM — MMRM includes treatment + baseline value + analysis visit + strata + analysis visit × treatment, where strata is the combination of randomization stratification factors; LS mean difference = -21.93, 95% CI 2-sided [-32.49 to -11.36]

10. Secondary Outcome: LS Mean Change From Baseline to Week 16 in Haptoglobin Level During the RCP
Description: as for outcome 3
Time Frame: Baseline and Week 16
Population: The ITT set included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
g/L | -0.02 (0.033) | 0.12 (0.063)
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.0369, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = -0.14, 95% CI 2-sided [-0.28 to -0.01]

11. Secondary Outcome: LS Mean Change From Baseline to Week 16 in Linear Analog Scale Assessment (LASA) Scores During the RCP
Description: The LASA consists of 3 items, where the respondents were asked to rate their perceived level of functioning. Specific domains included activity level, ability to carry out daily activities, and an item for overall QoL. Their level of functioning was reported on a 0 to 100 scale with 0 indicates "As low as could be" and 100 indicates "As high as could be". The combined score ranged from 0 to 300, with higher scores corresponding to a higher QoL.
Time Frame: Baseline and Week 16
Population: The ITT set included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
Score on a scale | 49.38 (10.189) | -9.72 (18.988)
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.0069, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = 59.10, 95% CI 2-sided [16.88 to 101.32]

12. Secondary Outcome: LS Mean Change From Baseline to Week 16 in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 Scale (QLQ-C30) Scores During the RCP
Description: The EORTC QLQ-C30 questionnaire (version 3.0) consists of 30 questions comprised of both multi-item scales and single-item measures to assess overall QoL in subjects. Questions are designated by functional scales, symptom scales, and global subject QoL/overall perceived health status. For the first 28 questions the 4 possible responses are "Not at all' (1), 'A little' (2), 'Quite a bit' (3) and 'Very much' (4). For the remaining 2 questions the response is requested on a 7-point scale from 1 ('Very poor') to 7 ('Excellent'). The raw scale scores were linear transformed, producing scale scores that ranged from 0% to 100%. A high scale score represents a higher response level. Hence for the functional scales and the global health status a higher score indicates a better QoL, whilst for the symptom scale scores this is implied by a lower score.
Time Frame: Baseline and Week 16
Population: The ITT set included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
Score on a scale
  Global Health Status/QoL | 15.91 (3.635) | -2.71 (8.515)
  Functional Scales - Physical functioning | 16.92 (2.081) | 4.06 (3.605)
  Functional Scales - Role functioning | 15.39 (3.930) | -9.04 (6.954)
  Functional Scales - Emotional functioning | 7.98 (3.366) | 3.86 (7.237)
  Functional Scales - Cognitive functioning | 5.76 (3.258) | -3.80 (6.420)
  Functional Scales - Social functioning | 15.08 (2.946) | 3.82 (6.349)
  Symptom Scales - Fatigue | -22.93 (3.321) | -2.18 (6.644)
  Symptom Scales - Nausea and vomiting | -0.34 (1.632) | -0.33 (3.876)
  Symptom Scales - Pain | -0.74 (4.323) | 2.01 (7.841)
  Symptom Scales - Dyspnoea | -20.12 (3.488) | -5.55 (7.019)
  Symptom Scales - Insomnia | -9.18 (3.955) | -9.50 (7.090)
  Symptom Scales - Appetite loss | -3.76 (3.357) | 4.19 (7.009)
  Symptom Scales - Constipation | 2.98 (3.248) | 1.19 (8.129)
  Symptom Scales - Diarrhoea | 0.31 (3.711) | 1.68 (8.204)
  Symptom Scales - Financial difficulties | -6.82 (3.853) | 0.58 (6.297)
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Global Health Status/QoL: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.0486, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = 18.62, 95% CI 2-sided [0.12 to 37.13]
Statistical Analysis 2: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Functional Scales - Physical functioning: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.0023, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = 12.86, 95% CI 2-sided [4.86 to 20.86]
Statistical Analysis 3: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Functional Scales - Role functioning: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.0027, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = 24.43, 95% CI 2-sided [8.84 to 40.01]
Statistical Analysis 4: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Functional Scales - Emotional functioning: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.6013, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = 4.11, 95% CI 2-sided [-11.58 to 19.80]
Statistical Analysis 5: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Functional Scales - Cognitive functioning: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.1792, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = 9.56, 95% CI 2-sided [-4.52 to 23.64]
Statistical Analysis 6: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Functional Scales - Social functioning: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.1039, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = 11.27, 95% CI 2-sided [-2.38 to 24.92]
Statistical Analysis 7: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Symptom Scales - Fatigue: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.0062, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = -20.74, 95% CI 2-sided [-35.29 to -6.19]
Statistical Analysis 8: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Symptom Scales - Nausea and vomiting: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.9975, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = -0.01, 95% CI 2-sided [-8.38 to 8.35]
Statistical Analysis 9: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Symptom Scales - Pain: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.7554, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = -2.76, 95% CI 2-sided [-20.36 to 14.85]
Statistical Analysis 10: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Symptom Scales - Dyspnoea: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.0620, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = -14.57, 95% CI 2-sided [-29.90 to 0.76]
Statistical Analysis 11: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Symptom Scales - Insomnia: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.9686, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = 0.32, 95% CI 2-sided [-15.67 to 16.30]
Statistical Analysis 12: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Symptom Scales - Appetite loss: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.3002, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = -7.95, 95% CI 2-sided [-23.23 to 7.33]
Statistical Analysis 13: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Symptom Scales - Constipation: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.8374, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = 1.79, 95% CI 2-sided [-15.70 to 19.29]
Statistical Analysis 14: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Symptom Scales - Diarrhoea: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.8775, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = -1.38, 95% CI 2-sided [-19.28 to 16.52]
Statistical Analysis 15: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Symptom Scales - Financial difficulties: Difference in LS mean; Test type: Other — [test comment as in outcome 9, analysis 1]; p = 0.3066, MMRM — [p-value comment as in outcome 9, analysis 1]; LS mean difference = -7.40, 95% CI 2-sided [-21.76 to 6.95]

13. Secondary Outcome: Total Number of PRBC Units Transfused During the RCP
Description: Subjects who withdrew during the RCP before Week 16 will have their number of units of PRBC estimated from the duration they were in the study.
Time Frame: Day 1 to Week 16
Population: The ITT set included all randomized subjects.
Measure: Number; unit: PRBC units
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 41 | 39
PRBC units | 26 | 198
Statistical Analysis 1: Comparison: Pegcetacoplan to Pegcetacoplan vs Eculizumab to Pegcetacoplan; Test type: Other — Wilcoxon rank-sum test P-value for the comparison between treatments is based on median using stratified non-parametric analysis. The 95% CI is constructed using Hodges-Lehmann Estimation of Location Shift; p < 0.0001, Wilcoxon rank-sum test; Median Difference (Final Values) = 3.0, 95% CI 2-sided [2.0 to 4.0]

14. Secondary Outcome: Mean Change From Baseline to Week 48 in Hb Level During the Treatment Period
Description: as for outcome 1
Time Frame: Baseline and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 33 | 30
g/dL | 2.47 (1.72) | 2.93 (2.09)

15. Secondary Outcome: Mean Change From Week 17 to Week 48 in Hb Level During the Open-label Period
Description: as for outcome 1
Time Frame: Week 17 and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Open-label Period: Continue Pegcetacoplan: On Day 1 of the RCP, the subjects were randomized to receive monotherapy with SC infusions of pegcetacoplan 1080 mg twice-weekly or every 3 days up to the end of the open-label period (Week 48).
- Open-label Period: Crossover to Pegcetacoplan: Subjects entered the open-label run-in period where they received pegcetacoplan 1080 mg twice-weekly in addition to eculizumab for 4 weeks (Week 17 to Week 20) before receiving monotherapy with SC infusions of pegcetacoplan 1080 mg twice-weekly or every 3 days up to the end of the open-label period (Week 48).
Arm/Group | Open-label Period: Continue Pegcetacoplan | Open-label Period: Crossover to Pegcetacoplan
Number analyzed (Participants) | 33 | 29
g/dL | -0.16 (1.154) | 2.89 (2.078)

16. Secondary Outcome: Mean Change From Baseline to Week 48 in ARC During the Treatment Period
Description: as for outcome 3
Time Frame: Baseline and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 31 | 29
10^9 cells/L | -135.64 (67.90) | -128.22 (59.60)

17. Secondary Outcome: Mean Change From Week 17 to Week 48 in ARC During the Open-label Period
Description: as for outcome 3
Time Frame: Week 17 and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Open-label Period: Continue Pegcetacoplan | Open-label Period: Crossover to Pegcetacoplan
Number analyzed (Participants) | 31 | 29
10^9 cells/L | -6.50 (26.471) | -121.15 (70.969)

18. Secondary Outcome: Mean Change From Baseline to Week 48 in LDH Level During the Treatment Period
Description: as for outcome 3
Time Frame: Baseline and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 33 | 30
U/L | -41.53 (153.68) | -105.27 (315.59)

19. Secondary Outcome: Mean Change From Week 17 to Week 48 in LDH Level During the Open-label Period
Description: as for outcome 3
Time Frame: Week 17 and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Open-label Period: Continue Pegcetacoplan | Open-label Period: Crossover to Pegcetacoplan
Number analyzed (Participants) | 33 | 28
U/L | 8.03 (129.285) | -46.84 (292.607)

20. Secondary Outcome: Mean Change From Baseline to Week 48 in FACIT-Fatigue Scale Score During the Treatment Period
Description: The FACIT-fatigue scale version 4 is a 13-item Likert scaled instrument where the subject was presented with 13 statements and asked to indicate their response as it applied to the past 7 days. The 5 possible responses were 'Not at all' (0), 'A little bit (1), 'Somewhat' (2), 'Quite a bit' (3) and 'Very much' (4). With 13 statements the total score had a range of 0 to 52. A higher score corresponds to a higher QoL. Baseline was the last available, nonmissing observation before taking the first dose of pegcetacoplan. Data collected after transfusion is excluded from analysis.
Time Frame: Baseline and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 30 | 29
Score on a scale | 10.14 (9.06) | 9.62 (10.34)

21. Secondary Outcome: Mean Change From Week 17 to Week 48 in FACIT-Fatigue Scale Score During the Open-label Period
Description: The FACIT-fatigue scale is a 13 item Likert scaled instrument where the subject was presented with 13 statements and asked to indicate their response as it applied to the past 7 days. The 5 possible responses were 'Not at all' (0), 'A little bit (1), 'Somewhat' (2), 'Quite a bit' (3) and 'Very much' (4). With 13 statements the total score had a range of 0 to 52. Higher score corresponds to a higher QoL.
Time Frame: Week 17 and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Open-label Period: Continue Pegcetacoplan | Open-label Period: Crossover to Pegcetacoplan
Number analyzed (Participants) | 30 | 26
Score on a scale | 1.28 (7.805) | 10.19 (10.973)

22. Secondary Outcome: Mean Change From Baseline to Week 48 in LASA Scores During the Treatment Period
Description: as for outcome 11
Time Frame: Baseline and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 29 | 29
Score on a scale | 58.66 (51.16) | 56.52 (65.55)

23. Secondary Outcome: Mean Change From Week 17 to Week 48 in LASA Scores During the Open-label Period
Description: as for outcome 21
Time Frame: Week 17 and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Open-label Period: Continue Pegcetacoplan | Open-label Period: Crossover to Pegcetacoplan
Number analyzed (Participants) | 30 | 26
Score on a scale | 13.13 (46.296) | 62.92 (60.053)

24. Secondary Outcome: Mean Change From Baseline to Week 48 in QLQ-C30 Scores During the Treatment Period
Description: The EORTC QLQ-C30 questionnaire (version 3.0) consists of 30 questions comprised of both multi-item scales and single-item measures to assess overall QoL in subjects. Questions are designated by functional scales, symptom scales, and global subject QoL/overall perceived health status. For the first 28 questions the 4 possible responses are 'Not at all' (1), 'A little' (2), 'Quite a bit' (3) and 'Very much' (4). For the remaining 2 questions the response is requested on a 7-point scale from 1 ('Very poor') to 7 ('Excellent'). The raw scale scores were linear transformed, producing scale scores that ranged from 0% to 100%. A high scale score represents a higher response level. Hence for the functional scales and the global health status a higher score indicates a better QoL, whilst for the symptom scale scores this is implied by a lower score.
Time Frame: Baseline and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pegcetacoplan to Pegcetacoplan | Eculizumab to Pegcetacoplan
Number analyzed (Participants) | 30 | 28
Score on a scale
  Global Health Status/QoL | 18.89 (17.635) | 13.99 (22.912)
  Functional Scales - Physical functioning | 15.33 (15.278) | 10.80 (17.765)
  Functional Scales - Role functioning | 16.67 (27.334) | 20.11 (27.595)
  Functional Scales - Emotional functioning | 10.28 (18.657) | 5.36 (17.005)
  Functional Scales - Cognitive functioning | 7.78 (23.462) | 0.00 (18.703)
  Functional Scales - Social functioning | 16.11 (24.166) | 14.88 (22.379)
  Symptom Scales - Fatigue | -21.48 (26.733) | -23.75 (29.506)
  Symptom Scales - Nausea and vomiting | -2.22 (11.357) | 0.00 (4.454)
  Symptom Scales - Pain | 0.56 (27.849) | 3.45 (20.596)
  Symptom Scales - Dyspnoea | -17.78 (29.985) | -27.59 (33.415)
  Symptom Scales - Insomnia | -6.67 (25.371) | 0.00 (28.172)
  Symptom Scales - Appetite loss | -7.78 (14.339) | -3.45 (22.440)
  Symptom Scales - Constipation | -1.11 (22.289) | -2.38 (8.742)
  Symptom Scales - Diarrhoea | 1.11 (29.664) | 5.95 (15.853)
  Symptom Scales - Financial difficulties | -15.56 (24.343) | -8.33 (19.510)

25. Secondary Outcome: Mean Change From Week 17 to Week 48 in QLQ-C30 Scores During the Open-label Period
Description: as for outcome 24
Time Frame: Week 17 and Week 48
Population: The ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Open-label Period: Continue Pegcetacoplan | Open-label Period: Crossover to Pegcetacoplan
Number analyzed (Participants) | 30 | 26
Score on a scale
  Global Health Status/QoL | 7.22 (19.664) | 23.08 (22.149)
  Functional Scales - Physical functioning | 0.89 (10.168) | 11.03 (17.173)
  Functional Scales - Role functioning | 5.00 (20.599) | 19.87 (22.617)
  Functional Scales - Emotional functioning | -2.22 (27.328) | 1.92 (13.806)
  Functional Scales - Cognitive functioning | -2.78 (16.999) | 2.56 (24.355)
  Functional Scales - Social functioning | 3.89 (18.919) | 12.18 (23.361)
  Symptom Scales - Fatigue | -2.96 (20.824) | -23.08 (28.790)
  Symptom Scales - Nausea and vomiting | -2.22 (5.762) | -4.49 (12.072)
  Symptom Scales - Pain | -2.78 (23.195) | -5.77 (21.051)
  Symptom Scales - Dyspnoea | 3.33 (25.295) | -19.23 (28.555)
  Symptom Scales - Insomnia | 8.89 (23.050) | -5.13 (27.797)
  Symptom Scales - Appetite loss | -8.89 (26.164) | -5.13 (22.494)
  Symptom Scales - Constipation | -1.11 (20.498) | -1.28 (11.473)
  Symptom Scales - Diarrhoea | -4.44 (28.679) | 3.85 (27.206)
  Symptom Scales - Financial difficulties | -2.22 (12.172) | -2.56 (16.119)

26. Secondary Outcome: Total Number of PRBC Units Transfused During the Open-Label Period
Description: Number of units of PRBC transfused to subjects in the open-label period are reported.
Time Frame: Week 17 to Week 48
Population: The ITT set included all randomized subjects.
Measure: Number; unit: PRBC Units
Groups:
- Open-label Run-in Period: Crossover to Pegcetacoplan: Subjects in the open-label run-in period received pegcetacoplan 1080 mg twice-weekly in addition to eculizumab for 4 weeks (Week 17 to Week 20).
Arm/Group | Open-label Period: Continue Pegcetacoplan | Open-label Period: Crossover to Pegcetacoplan | Open-label Run-in Period: Crossover to Pegcetacoplan
Number analyzed (Participants) | 38 | 39 | 38
PRBC Units | 68 | 110 | 14

ADVERSE EVENTS:
Time Frame: Day -28 to Week 54, a maximum of approximately 58 weeks
Groups:
- Run-in Period: Pegcetacoplan + Eculizumab: During the 4-week run-in period (Day -28 to ≤Day 1) all subjects received twice-weekly SC doses of pegcetacoplan 1080 mg in addition to their current dosage of eculizumab treatment. During the 4-week open-label run-in period (Week 17 to Week 20) subjects randomized to receive monotherapy with their pre-screening stable dose of eculizumab via intravenous infusion every 2 weeks during the RCP also received twice-weekly SC doses of pegcetacoplan 1080 mg.
- Open-label Period: Pegcetacoplan: The subjects who were randomized to receive monotherapy with SC infusions of pegcetacoplan 1080 mg twice-weekly or every 3 days during the RCP continued to receive monotherapy with pegcetacoplan until the end of the open-label period (Week 17 to Week 48). Subjects randomized to receive monotherapy with their pre-screening stable dose of eculizumab via intravenous infusion every 2 weeks during the RCP received monotherapy with SC infusions of pegcetacoplan 1080 mg twice-weekly or every 3 days after the open-label run-in period, up to the end of the open-label period (Week 20 to Week 48).
- RCP: Eculizumab: Subjects randomized to receive monotherapy with their pre-screening stable dose of eculizumab via intravenous infusion every 2 weeks during the RCP.
- RCP: Pegcetacoplan: Subjects randomized to receive monotherapy with SC infusions of pegcetacoplan 1080 mg twice-weekly or every 3 days during the RCP.
Arm/Group | Run-in Period: Pegcetacoplan + Eculizumab | Open-label Period: Pegcetacoplan | RCP: Eculizumab | RCP: Pegcetacoplan
All-Cause Mortality (participants affected / at risk) | 0/80 | 1/77 | 0/39 | 0/41
Serious Adverse Events (participants affected / at risk) | 4/80 | 18/77 | 5/39 | 7/41
Other Adverse Events (participants affected / at risk) | 71/80 | 71/77 | 36/39 | 36/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period: Pegcetacoplan + Eculizumab (N=80) | Open-label Period: Pegcetacoplan (N=77) | RCP: Eculizumab (N=39) | RCP: Pegcetacoplan (N=41)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to immunoglobulin therapy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 5 (5) | 1 (1) | 2 (2)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period: Pegcetacoplan + Eculizumab (N=80) | Open-label Period: Pegcetacoplan (N=77) | RCP: Eculizumab (N=39) | RCP: Pegcetacoplan (N=41)
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | 1 (1) | 3 (3)
Injection site erythema (General disorders) | 33 (75) | 9 (127) | 0 (0) | 7 (44)
Fatigue (General disorders) | 5 (5) | 8 (11) | 6 (7) | 2 (2)
Pyrexia (General disorders) | 6 (6) | 6 (9) | 1 (1) | 1 (1)
Injection site pruritus (General disorders) | 12 (14) | 5 (7) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 4 (4) | 5 (7) | 3 (3)
Injection site bruising (General disorders) | 2 (3) | 3 (7) | 0 (0) | 2 (2)
Injection site induration (General disorders) | 5 (12) | 5 (27) | 0 (0) | 3 (8)
Injection site reaction (General disorders) | 8 (26) | 2 (8) | 0 (0) | 4 (56)
Injection site swelling (General disorders) | 10 (18) | 1 (4) | 0 (0) | 4 (6)
Injection site pain (General disorders) | 6 (13) | 4 (68) | 0 (0) | 1 (9)
Vaccination site pain (General disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (5) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 13 (14) | 9 (14) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (5) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (9) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (4) | 1 (1)
Headache (Nervous system disorders) | 10 (12) | 8 (13) | 9 (10) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3) | 5 (5) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 11 (15) | 2 (2) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 2 (4) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 3 (3) | 2 (2) | 2 (3) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6) | 2 (2) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 4 (4) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 1 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 12 (13) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 7 (8) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 7 (7) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 6 (7) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT03500549/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT03500549/SAP_001.pdf